CLINICAL TRIAL: NCT05122416
Title: Optimization of Spleen VCTE Examinations with FibroScan
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Amendment has done in February 2024 in Spain to include patients with high BMI above 35 kg/m². It has been decided to terminate the patient inclusions earlier (after 33 patients) due to not reilable exams and no good quality examinations
Sponsor: Echosens (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: M139
Record Dates: First submitted 2021-11-03; First posted 2021-11-16 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Spleen; Fibrosis
Keywords: FibroScan; Vibration Control Transient Elastography; Spleen Stiffness Measurement
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Intervention Model Description: There will be 6 different groups of patients depending on the spleen to skin distance and the presence or absence of splenomegaly. Every patient in every group will do an ultrasound and 2 FibroScan exams. The differences between Group 1 (1a and 1b), Group 2 (2a and 2b) and Group 3 (3a and 3b) are the probes that will be used to do the FibroScan.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- Group 1a: SSD<15mm and with splenomegaly (Experimental): Patients with a Spleen to Skin Distance less than 15mm and who present a splenomegaly.
  Interventions: Device: FibroScan examination (S); Device: FibroScan examination (Standard M)
- Group 1b: SSD<15mm and without splenomegaly (Experimental): Patients with a Spleen to Skin Distance less than 15mm and who does not present a splenomegaly.
  Interventions: Device: FibroScan examination (S); Device: FibroScan examination (Standard M)
- Group 2a : 15<SSD<25mm and with splenomegaly (Experimental): Patients with a Spleen to Skin Distance between 15 and 25 mm and who present a splenomegaly.
  Interventions: Device: FibroScan examination (M); Device: FibroScan examination (Standard M)
- Group 2b : 15<SSD<25mm and without splenomegaly (Experimental): Patients with a Spleen to Skin Distance between 15 and 25 mm and who does not present a splenomegaly.
  Interventions: Device: FibroScan examination (M); Device: FibroScan examination (Standard M)
- Group 3.1.a: SSD≥25mm and with splenomegaly (Experimental): Patients with a Spleen to Skin Distance higher than 25 mm and who present a splenomegaly.
  Interventions: Device: FibroScan examination (XL); Device: FibroScan examination (Standard M)
- Group 3.1.b: SSD≥25mm and without splenomegaly (Experimental): Patients with a Spleen to Skin Distance higher than 25 mm and who does not present a splenomegaly.
  Interventions: Device: FibroScan examination (XL); Device: FibroScan examination (Standard M)
- 3.2 Patient with BMI >or = to 35kg/m² (Experimental): Patients with a Spleen to Skin Distance higher than 25 mm and BMI > or = to 35kg/m².
  Interventions: Device: FibroScan examination (M); Device: FibroScan examination (XL); Device: FibroScan examination (Standard M)

INTERVENTIONS:
Device: FibroScan examination (S) — A FibroScan examination with the Exploratory S probe.
  Arms: Group 1a: SSD<15mm and with splenomegaly; Group 1b: SSD<15mm and without splenomegaly
Device: FibroScan examination (M) — A FibroScan examination with the Optimized M probe.
  Arms: 3.2 Patient with BMI >or = to 35kg/m²; Group 2a : 15<SSD<25mm and with splenomegaly; Group 2b : 15<SSD<25mm and without splenomegaly
Device: FibroScan examination (XL) — A FibroScan examination with the Exploratory XL probe.
  Arms: 3.2 Patient with BMI >or = to 35kg/m²; Group 3.1.a: SSD≥25mm and with splenomegaly; Group 3.1.b: SSD≥25mm and without splenomegaly
Device: FibroScan examination (Standard M) — A FibroScan examination with the Standard M probe.

SUMMARY:
This is an European, prospective, interventional, and multicenter clinical investigation which main objective is to develop a spleen examination dedicated to overweight or obese patients and assess its applicability. It will take place in 4 sites (1 site in the Netherlands, 2 sites in Spain and 1 site in Romania) to include a total of 500 patients (adults and children).

ELIGIBILITY:
Inclusion Criteria:

1. Adult or pediatric patient able to give written informed consent (parents/legal tutors in case of minor patients),
2. Patient affiliated to the healthcare system
3. Adult or children patient followed for a liver disease a suspicion of liver disease or for a consequence of a liver disease, with or without splenomegaly and having a spleen to skin distance (SSD) measurement performed during the screening ultrasound exam.

Exclusion Criteria:

1. Vulnerable patient- other than pediatric patients
2. Patients with ascites

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 433 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-11-22 (Actual); Study Completion 2024-11-22 (Actual)

PRIMARY OUTCOMES:
Success rate of the spleen stiffness measurement (SSM) exam with both the optimized M+ probe and the exploratory XL+ probe, defined with at least 8 valid measurements after the exam quality control | At baseline visit
  The success rate is calculated with the number of valid measurements vs the total measurements done by the operator for every exam. The FibroScan will automatically analyze the measurement and based on some validity criteria will define the measurement as "valid" (will lead to a reliable SSM measurement) or "invalid" (will lead to a non-reliable SSM measurement).

SECONDARY OUTCOMES:
Success rate of the spleen stiffness measurement (SSM) exam with the S probe, defined with at least 8 valid measurements after the exam quality control. | At baseline visit
  The success rate is calculated with the number of valid measurements vs the total measurements done by the operator for every exam. The FibroScan will automatically analyze the measurement and based on some validity criteria will define the measurement as "valid" (will lead to a reliable SSM measurement) or "invalid" (will lead to a non-reliable SSM measurement).
Success rate of the spleen stiffness measurement (SSM) exam with the optimized M probe, defined with at least 8 valid measurements after the exam quality control. | At baseline visit
  The success rate is calculated with the number of valid measurements vs the total measurements done by the operator for every exam. The FibroScan will automatically analyze the measurement and based on some validity criteria will define the measurement as "valid" (will lead to a reliable SSM measurement) or "invalid" (will lead to a non-reliable SSM measurement).
Change of the applicability with the Spleen Targeting Tool (STT) and the automatic depth adaptation mode enabled. | At baseline visit
  This will be tested with unilateral Wilcoxon signed rank test comparing success rates with and without STT and with and without automatic depth adaptation.

CONTACTS AND LOCATIONS:
Overall Officials: Robert de Knegt, PhD, Principal Investigator — University Medical Center Rotterdam
Locations (4):
- University Medical Center Rotterdam, Rotterdam, Netherlands
- Regional Institute of Gastroenterology and Hepatology "Octavian Fodor" (IRGH), Cluj-Napoca, Romania
- Spain (2):
  - Hospital Puerta de Hierro Majadahonda, Madrid
  - Hospital Universitario La Paz, Madrid